CLINICAL TRIAL: NCT01451749
Title: Phase III Study of Shenwu Capsule in Treating Amnestic Mild Cognitive Impairment
Brief Title: Efficacy and Safety Study of Shenwu Capsule
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: North China Pharmaceutical Group Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFDA2001ZL116-SW; NorthChinaPGC (Other: State Adminstration of Food and Drug of China)
Record Dates: First submitted 2011-10-11; First posted 2011-10-14 (Estimated); Results first posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — shenwu; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shenwu Capsule (Experimental): Shenwu Capsule:1 capsule contains 451 mg of Shenwu extracts. 5 capsules/time, 3 times/day for 6 months.
  Placebo: Placebo identical to donepezil tablets,1 placebo tablet/time, 1 time/day for 6 months.
  Interventions: Drug: Shenwu Capsule
- Donepezil (Active Comparator): Donepezil: 1 tablet contains 5 mg of donepezil, 1 tablet/time, 1time/day for 6 months.
  Placebo: Placebo identical to shenwu capsules,5 placebo capsules/time,3 times/day for 6 months
  Interventions: Drug: Donepezil

INTERVENTIONS:
Drug: Shenwu Capsule — 1 shenwu capsule contains 451 mg extract from herbs.5 capsules/time, 3 times/day for 6 months.
  Placebo identified to donepezil: 1 tablet per time, 1 time per day for 6 months.
  Other Names: Shenwu
  Arms: Shenwu Capsule
Drug: Donepezil — This active drug is donepezil 5 mg tablet. 1 tablet/time, 1 time/day for 6 months.
  Placebo identical to shenwu capsules,5 capsules/time,3times/day for 6months.
  Other Names: Aricept
  Arms: Donepezil

SUMMARY:
The purpose of this phase III study is to further evaluate the effects of shenwu capsule, a traditional Chinese herbal medicine, on cognition, function and memory in patients with amnestic mild cognitive impairment (MCI) who are at greater risk for developing Alzheimer's disease, in a 6-month supervised protocol of a traditional Chinese herbal medicine. The results of this study may provide support for a relatively simple and inexpensive treatment strategy with herbal therapy that specifically targets individuals with the mild cognitive impairment that directly influence risk of developing dementia for older adults.

DETAILED DESCRIPTION:
Mild cognitive impairment (MCI) refers to a group of individuals who have some cognitive impairment but of insufficient severity to constitute dementia1,which is a transitional stage between normal aging and dementia. Amnestic MCI is the most common subtype of MCI, which shows the least reversion to normal, and is defined as a significant impairment in memory but with no impairment in activities of daily living. In an interventional study of patients meeting Petersen criteria for amnestic MCI, 16% progressed to dementia per year, 99% of whom received an AD diagnosis. Hence, MCI, in particular amnestic MCI is generally recognized in many cases to represent prodromal AD and becomes a new target for prevention and treatment of AD.

The specific aims for the study is to evaluate change in Efficacy and safety of shenwu capsule in treating amnestic MCI. Using a randomized controlled parallel group design, 324 older adults diagnosed with amnestic MCI participate in a 6-month supervised protocol of either shenwu capsule or donepezil. Cognitive testing and blood collection will occur at baseline, and months 3 and 6. Before the 6-month intervention, medial temporal atrophy (MTA) or hippocampal volume atrophy on the CT or MRI scan are assessed for all subjects. The results of this study may provide support for a safer and inexpensive treatment strategy that specifically targets individuals with the mild cognitive impairment that directly influence risk of developing dementia for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Chinese-speaking adults at least 55 to 80 years of age old, weighting between 45 to 90 kilograms, living in the community.
* diagnosed with amnestic MCI at screening: (1) memory complaint, corroborated by an informant; (2) abnormal memory function, as screened by the WMS-R Logical Memory II Delayed Story Recall subtest score <10.4 for age; (3) normal general cognitive function, as determined by a clinician's judgment based on a structured interview with the patients (MMSE of 24 to 30 score for education ); (4) no or minimal impairment in activities of daily living, as determined by a clinical interview with the patient and informant (IADL <16 score); and (5) not sufficiently impaired, cognitively and functionally, to meet NINCDS-ADRDA criteria for AD, as judged by an experienced AD research clinician. In addition, they were judged to be at stage 2-3 of the GDS, and to have a score of ≤12 of the HAMD for 17 items, of ≤4 on the HIS, and no or minimal medial temporal atrophy (MTA) or hippocampal volume atrophy on the MRI scan.
* The subjects required adequate vision and hearing to participate in study assessments. Patients receiving chronic aspirin therapy for cardio-protection (≤100 mg per day) or stable doses of antidepressants for at least 3 months were also eligible.

Exclusion Criteria:

* Significant neurologic disease that might affect cognition, such as a diagnosis of Alzheimer's disease, stroke, Parkinson's disease, multiple sclerosis, or severe head injury with loss of consciousness; a score of MMSE<24,or any major psychiatric disorder (e.g., DSM-IV-defined psychosis, major depression, bipolar disorder, or alcohol or substance abuse);
* Recent history of chronic use of NSAIDs or aspirin (>100 mg per day);
* History of upper gastrointestinal bleeding that required transfusion or surgery within the previous 3 years,or documented evidence of an active gastric or duodenal ulcer within the previous 3 months,or history of NSAID-associated ulcers;
* History of active malignancy except for basal cell carcinoma or squamous cell carcinoma of the skin, or prostate cancer, within the preceding 24 months;
* A chronic or acute renal, hepatic, or metabolic disorder; and uncontrolled hypertension and diabetes mellitus;
* History of hypersensitivity to the treatment drugs; or concomitant drugs (including anticonvulsant agents, anti-parkinsonian agents, antipsychotics, anxiolytics, hypnotic agents, neuroleptic agents, cholinomimetic agents, vitamin E, or ginkgo biloba extract or any other drugs including traditional Chinese herbal medicines which can affect memory); or participants in other clinical studies within the past 30 days.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2008-09; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinzhou Tian, MD,PhD, Study Chair — Dongzhimen Hospital, Beijing
Locations (1):
- Dongzhimen Hospital,BUCM, Beijing, China

REFERENCES:
- [Derived] Tian J, Shi J, Li T, Li L, Wang Z, Li X, Lv Z, Zheng Q, Wei M, Wang Y. Efficacy and Safety of an Herbal Therapy in Patients with Amnestic Mild Cognitive Impairment: A 24-Week Randomized Phase III Trial. Evid Based Complement Alternat Med. 2017;2017:4251747. doi: 10.1155/2017/4251747. Epub 2017 May 17. PMID 28596794

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 9 sites in China were conducted patients from September 1, 2008, to May 3, 2010.The 9 sites was medical clinic in hospital.
Groups:
- Shenwu Capsule: Shenwu Capsule: 1 shenwu capsule contains 451 mg extract from herbs. 5 capsules/time, 3 times/day for 6 months. Placebo identical to donepezil: 1 placebo tablet/time,1 time/day for 6 months
- Donepezil: Donepezil: This active drug is donepezil 5 mg tablet. 1 tablet/time, 1 time/day for 6 months.
  Placebo identical to shenwu capsules: 5 capsules/time,3times/day for 6months.
Period: Overall Study
Arm/Group | Shenwu Capsule | Donepezil
Started | 216 | 108
Completed | 184 | 94
Not Completed | 32 | 14
Not completed — Protocol Violation | 14 | 7
Not completed — Lost to Follow-up | 15 | 5
Not completed — Meet the exclusion criteria,and | 1 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: 216 in Shenwu capusle, and 108 in the Donepezil group was enrolled at baseline, 1 subjects in both group did not meet the inclusion criteria ,and 215 in Shenwu Capsule, and 107 in Donepezil were used to baseline analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Shenwu Capsule | Donepezil | Total
Number analyzed (Participants) | 215 | 107 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.67 (7.96) | 63.80 (8.25) | 62.97 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 61 | 188
  Male | 88 | 46 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 215 | 107 | 322
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 215 | 107 | 322
Mini-mental state examinition [Mean (Full Range); unit: units on a scale] — The Mini-mental State Examination(MMSE) is a brief 30-point questionnaire test that is used to screen for cognitive impairment. It is used to estimate the severity of cognitive impairment and to follow the course of cognitive changes in an individual over time, thus making it an effective way to document an individual's response to treatment. The scores of the MMSE ranges from 0 to 30, and a lower score indicate higher impairment. The MMSE score ranges from 24-30 points in both group.
  units on a scale | 27.38 [24 to 30] | 27.11 [24 to 30] | 27.30 [24 to 30]
Education [Number; unit: participants]
  Primary school | 40 | 26 | 66
  Longer than middle school | 175 | 81 | 256
Global Deterioration Scale [Number; unit: participants] — The Global Deterioration Scale (GDS), provides caregivers an overview of the stages of cognitive function for those suffering from a primary degenerative dementia such as Alzheimer's disease. It is broken down into 7 different stages. Stages 1-3 are the pre-dementia stages. Stages 4-7 are the dementia stages.
  Beginning in stage 5, an individual can no longer survive without assistance.
  participants
    Stage 1 | 0 | 1 | 1
    Stage 2 | 101 | 47 | 148
    Stage 3 | 114 | 59 | 173
Hamilton depression rating scale [Mean (Full Range); unit: units on a scale] — The Hamilton Rating Scale for Depression is designed for adults and is used to rate the severity of their depression by probing mood, feelings of guilt, suicide ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms.The HAMD scale contains 17 tems, each item is scored on a 3 or 5 point scale, and the total score is compared to the corresponding descriptor. The total score ranges from 0-52 points. A score of 0-7 is considered to be normal. Scores of 20 or higher indicate moderate, severe, or very severe depression. Both group ranges form 0-12 points.
  units on a scale | 6.44 [0 to 12] | 6.39 [0 to 12] | 6.40 [0 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Scores: Alzheimer Disease Assessment Scale-cognitive. Subscale (ADAS-cog)
Description: Cognition was assessed with the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) , at baseline (day 1 clinic visit) and at 12-week intervals thereafter until week 24. The ADAS-cog was designed specifically to evaluate the severity of cognitive dysfunctions characteristic of AD patients and includes 11 items. Among these items, memory, orientation, language function, practical ability, and attention are evaluated. The score on the ADAS-cog range from 0 to 70 point, with 0 point indicating no impairment and 70 points indicating severe impairment of cognition. In the Shenwu capsule group, the ADAS-cog score is ranges 3-38.3 points, and 3.3-30.7 points in the Donepezil group. The Change in cognitive scores was calculated as24 week minus the baseline.
Time Frame: baseline and 24 weeks
Population: the analyses for efficacy were conducted in the intent-to-treat population (ITT). The intent-to-treat population (ITT) consist all randomized population who take at least one dose of medication and at least one primary efficacy evaluation on treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Shenwu Capsule | Donepezil
Number analyzed (Participants) | 215 | 107
units on a scale | -4.23 [-4.71 to -3.75] | -4.31 [-4.99 to -3.63]

2. Secondary Outcome: Change in Memory Scores: The Delayed Story Recall (DSR) Test From the Adult Memory and Information Processing Battery (AMIPB)
Description: memory function was evaluated with the DSR subtest,at baseline (day 1 clinic visit), at the mid-study (week 12), and at the endpoint of treatment (week 24). The DSR is a tool which was designed to assess immediate registration of verbal information and retention over time. It contains six sub-tests: two verbal memory tests (one of which is a story recall), two visual memory tests and two information-processing tests. The story recall test includes immediate story recall (ISR) and delayed story recall (DSR). The DSR total score ranges from 0-56 points. Lowers score means higher impairment of memory.The Change in cognitive scores was calculated as 24 week minus the baseline.
Time Frame: Baseline and 24 weeks
Population: The efficacy measurement was conducted of ITT patients. The intent-to-treat population (ITT) consist all randomized population who take at least one dose of medication and at least one primary efficacy evaluation on treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Shenwu Capsule: 1 capsule contains 451 mg of Shenwu extracts. 5 capsules/time, 3 times/day for 6 months.
  Shenwu Capsule: 1 shenwu capsule contains 451 mg extract from herbs. 5 capsules/time, 3 times/day for 6 months. Placebo identical to donepezil: 1 placebo tablet/time,1 time/day for 6 months
- Donepezil: 1 tablet contains 5 mg of donepezil, 1 tablet/time, 1time/day for 6 months.
  Donepezil: This active drug is donepezil 5 mg tablet. 1 tablet/time, 1 time/day for 6 months.
  Placebo identical to shenwu capsules: 5 capsules/time,3times/day for 6months.
Arm/Group | Shenwu Capsule | Donepezil
Number analyzed (Participants) | 215 | 107
units on a scale | 9.45 [8.5 to 10.4] | 9.9 [8.49 to 11.34]

3. Secondary Outcome: Change in Functional Scores: Instrumental Activities of Daily Living (IADL).
Description: Functional ability was evaluated with the Instrumental Activities of Daily Living (IADL) IADL, at baseline (day 1 clinic visit), at the mid-study (week 12), and at the endpoint of treatment (week 24). The IADL contains eight items, which are the ability to use a telephone, shop, prepare food, run laundry, use modes of transportation, take responsibility for one's own medications, complete housekeeping, and handle finances,each items ranges from 1 to 4 points, 1 points means no problem, and 4 points means greater impairment in instumental acvtiveity of daily living.The total is sub of the eight items, and the total range of the IADL is 8-32 points, higher scores indicate greater impairments. The changes was calculted by weeks 24 minus baseline.
Time Frame: Baseline to weeks 24
Population: The efficacy measurement were conducted in the intent-to-treat population, the ITT consist all randomized population who take at least one dose of medication and at least one primary efficacy evaluation on treatment.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Shenwu Capsule | Donepezil
Number analyzed (Participants) | 215 | 107
units on a scale | 0.96 [0.75 to 1.18] | 1.18 [0.85 to 1.50]

ADVERSE EVENTS:
Time Frame: Baseline to weeks 24
Arm/Group | Shenwu Capsule | Donepezil
Serious Adverse Events (participants affected / at risk) | 0/216 | 0/108
Other Adverse Events (participants affected / at risk) | 39/216 | 62/108
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Shenwu Capsule (N=216) | Donepezil (N=108)
Insomnia or abnormal dreams (Nervous system disorders) | 5 | 18
Nausea (Gastrointestinal disorders) | 5 | 18
Abnormalalanine aminotransferas (ALT) (Hepatobiliary disorders) | 1 | 1
Skin rash (Skin and subcutaneous tissue disorders) | 0 | 1
Vomit (Gastrointestinal disorders) | 0 | 5
Diarrhea (Gastrointestinal disorders) | 0 | 14
Thirsty (General disorders) | 14 | 5
Sore throat (General disorders) | 9 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 5 | 0

LIMITATIONS AND CAVEATS:
First, there was no placebo group. As all subjects knew that they were being treated with one of two drugs, and all of the individuals who assessed the patients knew this as well, the results may have been influenced by a positive response bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less